CLINICAL TRIAL: NCT00758082
Title: Reinforcement of the Impact of a Functional Insulin Therapy Training Course by Telemonotoring With a PDA-phone in Type 1 Diabetic Patients. The TELFIT Study
Brief Title: Reinforcement of the Impact of a Functional Insulin Therapy Training Course by Telemonotoring With a PDA-phone in Type 1 Diabetic Patients. The TELFIT Study Patients
Acronym: TELFIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: AGIR à Dom (Other)
Responsible Party: Pr Pierre-Yves Benhamou, University Hospital Grenoble
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-A00389-46
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Last update posted 2010-03-11 (Estimated); Status verified 2010-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes; PDA phone (Personal Digital Assistant); HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients will have face to face visits at 3 months and no PDA-phone. Patients will record glycemia on paper support
  Interventions: Device: paper support
- 2 (Experimental): PDA-phone + phone consultations + standard visit at 3 months
  Interventions: Device: PDA-phone + telemonitoring

INTERVENTIONS:
Device: paper support — Patients will have face to face visits at 3 months and no PDA-phone. Patients will record glycemia on paper support.
  Arms: 1
Device: PDA-phone + telemonitoring — Patients will received PDA-phone + a telephone follow up + standard visit at 3 months
  Arms: 2

SUMMARY:
TELFIT is a monocenter, controlled, randomised trial. It focuses on type 1 diabetes patients that have attended a functional insulin therapy training course. The Primary objective of the TELFIT study is to evaluate whether a PDA with telemonitoring by phone reinforces the effects of the functional insulin therapy training course as compared with conventional care.

Main judgment criteria: comparison of HbA1c means between M0 (start) and M3(3 months)

DETAILED DESCRIPTION:
All patients will attend a functional insulin therapy training course and be randomized into 2 groups. One group will receive a PDA-phone and one month of phone consultations with a nurse and a physician. The other group will only have the usual paper support. This study compares the evolution of HbA1c in the 2 groups over a period of 3 months. It also assesses time spent by nurses and physicians, changes in quality of life, hypoglycaemia frequency and weight changes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for ≥ 6 months or more
* Age > 18 year old
* The patient has attended a functional insulin therapy class or workshop
* Insulin basal-bolus therapy for at least 6 months. At inclusion, patients should be treated either with a long-acting insulin and insulin rapid analog before each meal, or with rapid insulin analog delivered with a pump
* Ability to understand how the PDA-phone works and ability to use it
* Social Security membership or benefit from Social Security
* Patients equipped with a memory blood glucose monitor
* Informed consent, with a signed and approved form

Exclusion Criteria:

* Underage patient, major patient under guardianship or protected by the Law
* Patient with any unstable associated evolutive pathology that could cause a diabetes imbalance within the coming year
* Change in diabetes treatment within the 3 months before inclusion or planned during the study
* Patient who needs a more frequent diabetic follow-up than in the protocol (especially severe or evolving complication due to diabetes)
* Patient attending another education program within the 3 months before inclusion or planning to attend one during the study
* Patient with toxicomania, alcoholism or psychological troubles that could impact the study
* Type-2-diabetic patient
* Patient who doesn't need strict metabolic objectives
* Pregnant or possibly pregnant woman
* Person with no freedom (prisoner)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Comparison of HbA1c means | M0 (start) and M3 (3 months)

SECONDARY OUTCOMES:
Difference between theoretical insulin dose and actual dose, one week before the 3-month reevaluation session | M0 (start) and M3 (3 months)
DHP scale of quality of life and satisfaction dimension of the DQOL questionnaire | M0 (start) and M3 (3 months)
Time spent by physicians and nurses in the different groups | M0 (start) and M3 (3 months)
Weight changes during the 3-month period | M0 (start) and M3 (3 months)
Number of hypoglycemias (moderate and severe) during the 3-month period | M0 (start) and M3 (3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Y Benhamou, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France